CLINICAL TRIAL: NCT01927302
Title: The Center for the Neurobiology of Language Recovery (CNLR)
Brief Title: Neurobiology of Language Recovery in Aphasia: Natural History and Treatment-Induced Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Cynthia K Thompson, Ralph and Jean Sundin Professor of Communication Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P50; P50DC012283 (NIH)
Record Dates: First submitted 2013-07-29; First posted 2013-08-22 (Estimated); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Aphasia; Dysgraphia; Anomia; Agrammatism; Stroke
Keywords: Aphasia; Dysgraphia; Anomia; Agrammatism; Stroke; Language Recovery; Treatment; Biomarkers of Recovery
MeSH Terms: conditions — Aphasia; Agraphia; Anomia; Aphasia, Broca; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Naming Deficits (Experimental): Language treatment will focus on improving naming deficits in people who have aphasia. An experimental group will receive treatment focusing on naming objects and a control/natural history group will receive no treatment. Both groups will be assessed at baseline (week 0), at week 12, and at week 24.
  Interventions: Behavioral: Treatment Focusing on Naming Objects; Behavioral: No Treatment
- Spelling and/or Writing Deficits (Experimental): Language treatment will focus on improving writing and/or spelling deficits in people who have aphasia. An experimental group will receive treatment focusing on improving spelling abilities and a control/natural history group will receive no treatment. Both groups will be assessed at baseline (week 0), at week 12, and at week 24.
  Interventions: Behavioral: Treatment Focusing on Improving Spelling Abilities; Behavioral: No Treatment
- Sentence Processing (Experimental): Language treatment will focus on improving sentence comprehension and production deficits in people who have aphasia. An experimental group will receive treatment focusing on improving sentence processing and a control/natural history group will receive no treatment. Both groups will be assessed at baseline (week 0), at week 12, and at week 24.
  Interventions: Behavioral: Treatment Focusing on Improving Sentence Processing; Behavioral: No Treatment

INTERVENTIONS:
Behavioral: Treatment Focusing on Naming Objects — Treatment will be administered from week 0 until week 12.
  Other Names: Language treatment
  Arms: Naming Deficits
Behavioral: Treatment Focusing on Improving Spelling Abilities — Treatment will be administered from week 0 until week 12.
  Other Names: Language Treatment
  Arms: Spelling and/or Writing Deficits
Behavioral: Treatment Focusing on Improving Sentence Processing — Treatment will be administered from week 0 until week 12.
  Other Names: Language Treatment
  Arms: Sentence Processing
Behavioral: No Treatment — No treatment will be administered.

SUMMARY:
The purpose of this study is to investigate the effects of treatment for specific language deficits in people with aphasia. In addition to language and cognitive measures, changes in brain function will also be gathered before and after the treatment is administered in order to track any changes resulting from receiving treatment.

DETAILED DESCRIPTION:
Naming Impairments (Anomia):

The labs of Dr. Swathi Kiran (Boston University) and Dr. David Caplan (Harvard University, Massachusetts General Hospital) will be studying language recovery in adults with anomia (naming impairments) following a stroke. Participants will receive treatment focusing on the semantic features of common objects (e.g., that birds can fly). The study will examine how naming and other language abilities change in response to treatment, as well as how the brain changes, as measured by magnetic resonance imaging (MRI) and other techniques.

Spelling/Writing Impairments (Dysgraphia):

At Johns Hopkins University, the lab of Dr. Brenda Rapp will investigate the neurobiology of language recovery in individuals with dysgraphia (spelling/writing impairments) resulting from a stroke. In this study, treatment will focus on improving spelling ability. The study will examine how spelling and other language abilities change in response to treatment, as well as how the brain changes, as measured by magnetic resonance imaging (MRI) and other techniques.

Deficits in Sentence Comprehension & Production:

Dr. Cynthia Thompson's lab at Northwestern University will investigate language recovery in individuals with deficits in sentence production and comprehension. Treatment focuses on production and comprehension of complex sentences. At baseline (week 0) and after the treatment period (at week 12), participants take part in language, eye-tracking, and MRI testing, in order to learn how the processing of language, as well as brain function, changes as a result of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aphasia following a stroke
* Stoke was at least 1 year ago
* Medically stable
* Right-handed
* Normal or 'corrected to normal' vision and hearing
* English as primary language
* At least a high school education

Exclusion Criteria:

* History of neurological disease, head trauma, psychiatric disorders, alcoholism, or developmental speech, language, or learning disabilities

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Change in language and cognitive abilities as a result of treatment | week 0 to week 12
  Standard and non-standard measures of language and cognitive abilities will be gathered at baseline (week 0) to see if language deficits improve after treatment is administered (week 12).

SECONDARY OUTCOMES:
Composite change in brain function as a result of treatment | week 0 to week 12
  Neural correlates of treatment effects will be examined using:
  * Functional Magnetic Resonance Imaging (fMRI)
  * Diffusion Tensor Imaging (DTI)
  * Perfusion Imaging
  * Functional Connectivity
  * Rest state Connectivity
Maintenance of language and cognitive abilities as a result of treatment | week 12 to week 24
  Standard and non-standard measures of language and cognitive abilities administered at week 12 will be compared to those administered at week 24 to see if improvement in language abilities as a result of treatment is maintained.
Maintenance of composite changes in brain function as a result of treatment | week 12 to week 24
  Neural correlates of treatment effects that are maintained for 12 weeks after treatment ends (week 12 to week 24) will be examined using:
  * Functional Magnetic Resonance Imaging (fMRI)
  * Diffusion Tensor Imaging (DTI)
  * Perfusion Imaging
  * Functional Connectivity
  * Rest state Connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia K Thompson, PhD, Study Director — Northwestern University; David Caplan, MDCM, PhD, Principal Investigator — Harvard University Massachusetts General Hospital; Brenda Rapp, PhD, Principal Investigator — Johns Hopkins University; Swathi Kiran, PhD, CCC-SLP, Principal Investigator — Boston University; Todd B Parrish, PhD, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - Harvard University, Cambridge, Massachusetts

REFERENCES:
- [Background] Walenski M, Europa E, Caplan D, Thompson CK. Neural networks for sentence comprehension and production: An ALE-based meta-analysis of neuroimaging studies. Hum Brain Mapp. 2019 Jun 1;40(8):2275-2304. doi: 10.1002/hbm.24523. Epub 2019 Jan 28. PMID 30689268
- [Background] Kiran S, Thompson CK. Neuroplasticity of Language Networks in Aphasia: Advances, Updates, and Future Challenges. Front Neurol. 2019 Apr 2;10:295. doi: 10.3389/fneur.2019.00295. eCollection 2019. PMID 31001187
- [Background] Crinion J, Holland AL, Copland DA, Thompson CK, Hillis AE. Neuroimaging in aphasia treatment research: quantifying brain lesions after stroke. Neuroimage. 2013 Jun;73:208-14. doi: 10.1016/j.neuroimage.2012.07.044. Epub 2012 Jul 27. PMID 22846659
- [Background] Kiran S, Ansaldo A, Bastiaanse R, Cherney LR, Howard D, Faroqi-Shah Y, Meinzer M, Thompson CK. Neuroimaging in aphasia treatment research: standards for establishing the effects of treatment. Neuroimage. 2013 Aug 1;76:428-35. doi: 10.1016/j.neuroimage.2012.10.011. Epub 2012 Oct 9. PMID 23063559
- [Background] Meinzer M, Beeson PM, Cappa S, Crinion J, Kiran S, Saur D, Parrish T, Crosson B, Thompson CK; Neuroimaging in Aphasia Treatment Research Workshop. Neuroimaging in aphasia treatment research: consensus and practical guidelines for data analysis. Neuroimage. 2013 Jun;73:215-24. doi: 10.1016/j.neuroimage.2012.02.058. Epub 2012 Feb 24. PMID 22387474
- [Background] Rapp B, Caplan D, Edwards S, Visch-Brink E, Thompson CK. Neuroimaging in aphasia treatment research: issues of experimental design for relating cognitive to neural changes. Neuroimage. 2013 Jun;73:200-7. doi: 10.1016/j.neuroimage.2012.09.007. Epub 2012 Sep 10. PMID 22974976
- [Background] Ditges R, Barbieri E, Thompson CK, Weintraub S, Weiller C, Mesulam MM, Kummerer D, Schroter N, Musso M. German Language Adaptation of the NAVS (NAVS-G) and of the NAT (NAT-G): Testing Grammar in Aphasia. Brain Sci. 2021 Apr 8;11(4):474. doi: 10.3390/brainsci11040474. PMID 33918022
- [Background] Thompson CK. Neurocognitive Recovery of Sentence Processing in Aphasia. J Speech Lang Hear Res. 2019 Nov 22;62(11):3947-3972. doi: 10.1044/2019_JSLHR-L-RSNP-19-0219. Epub 2019 Nov 22. PMID 31756151
- [Background] Schuchard J, Thompson CK. Implicit and explicit learning in individuals with agrammatic aphasia. J Psycholinguist Res. 2014 Jun;43(3):209-24. doi: 10.1007/s10936-013-9248-4. PMID 23532578
- [Background] Wang H, Yoshida M, Thompson CK. Parallel functional category deficits in clauses and nominal phrases: The case of English agrammatism. J Neurolinguistics. 2014 Jan;27(1):75-102. doi: 10.1016/j.jneuroling.2013.09.001. PMID 26379370
- [Background] Thompson CK, Faroqi-Shah Y, & Lee J. (2015). Models of sentence production. In: A. Hillis (Ed.). The handbook of adult language disorders: Integrating cognitive neuropsychology, neurology, and rehabilitation. Second Edition (pp. 328-354). New York: Psychology Press.
- [Background] Thompson CK, Kielar A. (2014). Neural bases of sentence processing: evidence from neurolinguistic and neuroimaging studies. In M. Goldrick, V. Ferreira, & M. Miozzo (Eds.) The Oxford Handbook of Language Production (pp. 47-69). New York: Oxford University Press.
- [Background] Thompson CK, Meltzer-Asscher, A. (2014). Neurocognitive mechanisms of verb argument structure processing. In Asaf Bachrach, Isabelle Roy and Linaea Stockall (Eds.) Structuring the Argument: Multidisciplinary research on verb argument structure (pp. 141-168). John Benjamins.
- [Background] Iorga M, Higgins J, Caplan D, Zinbarg R, Kiran S, Thompson CK, Rapp B, Parrish TB. Predicting language recovery in post-stroke aphasia using behavior and functional MRI. Sci Rep. 2021 Apr 19;11(1):8419. doi: 10.1038/s41598-021-88022-z. PMID 33875733
- [Background] Ingo C, Sui Y, Chen Y, Parrish TB, Webb AG, Ronen I. Parsimonious continuous time random walk models and kurtosis for diffusion in magnetic resonance of biological tissue. Front Phys. 2015 Mar;3:11. doi: 10.3389/fphy.2015.00011. Epub 2015 Mar 16. PMID 28344972
- [Background] Alpert K, Kogan A, Parrish T, Marcus D, Wang L. The Northwestern University Neuroimaging Data Archive (NUNDA). Neuroimage. 2016 Jan 1;124(Pt B):1131-1136. doi: 10.1016/j.neuroimage.2015.05.060. Epub 2015 May 30. PMID 26032888
- [Background] Ingo C, Magin RL, Parrish TB. New Insights into the Fractional Order Diffusion Equation Using Entropy and Kurtosis. Entropy (Basel). 2014 Nov;16(11):5838-5852. doi: 10.3390/e16115838. Epub 2014 Nov 6. PMID 28344436
- [Background] Meier EL, Johnson JP, Pan Y, Kiran S. The utility of lesion classification in predicting language and treatment outcomes in chronic stroke-induced aphasia. Brain Imaging Behav. 2019 Dec;13(6):1510-1525. doi: 10.1007/s11682-019-00118-3. PMID 31093842
- [Background] Gilmore N, Meier EL, Johnson JP, Kiran S. Nonlinguistic Cognitive Factors Predict Treatment-Induced Recovery in Chronic Poststroke Aphasia. Arch Phys Med Rehabil. 2019 Jul;100(7):1251-1258. doi: 10.1016/j.apmr.2018.12.024. Epub 2019 Jan 9. PMID 30639272
- [Background] Gilmore N, Meier EL, Johnson JP, Kiran S. Typicality-based semantic treatment for anomia results in multiple levels of generalisation. Neuropsychol Rehabil. 2020 Jun;30(5):802-828. doi: 10.1080/09602011.2018.1499533. Epub 2018 Jul 20. PMID 30027828
- [Background] Meier EL, Johnson JP, Kiran S. Left frontotemporal effective connectivity during semantic feature judgments in patients with chronic aphasia and age-matched healthy controls. Cortex. 2018 Nov;108:173-192. doi: 10.1016/j.cortex.2018.08.006. Epub 2018 Aug 27. PMID 30243049
- [Background] Meier EL, Johnson JP, Villard S, Kiran S. Does Naming Therapy Make Ordering in a Restaurant Easier? Dynamics of Co-Occurring Change in Cognitive-Linguistic and Functional Communication Skills in Aphasia. Am J Speech Lang Pathol. 2017 May 17;26(2):266-280. doi: 10.1044/2016_AJSLP-16-0028. PMID 28196373
- [Background] Meier EL, Kapse KJ, Kiran S. The Relationship between Frontotemporal Effective Connectivity during Picture Naming, Behavior, and Preserved Cortical Tissue in Chronic Aphasia. Front Hum Neurosci. 2016 Mar 16;10:109. doi: 10.3389/fnhum.2016.00109. eCollection 2016. PMID 27014039
- [Background] Meier EL, Lo M, Kiran S. Understanding semantic and phonological processing deficits in adults with aphasia: Effects of category and typicality. Aphasiology. 2016;30(6):719-749. doi: 10.1080/02687038.2015.1081137. Epub 2015 Sep 12. PMID 27041784
- [Background] Kiran S, Meier EL, Kapse KJ, Glynn PA. Changes in task-based effective connectivity in language networks following rehabilitation in post-stroke patients with aphasia. Front Hum Neurosci. 2015 Jun 9;9:316. doi: 10.3389/fnhum.2015.00316. eCollection 2015. PMID 26106314
- [Background] Vallila-Rohter S, Kiran S. (2015). Diagnosis and Treatment of Semantic Impairments. In A. Hillis (Ed.) Handbook on Adult Language Disorders. Taylor & Francis/Psychology Press of 711 Third Avenue, 8th Floor, New York, NY 10017.
- [Background] Breining B, Rapp B. Investigating the mechanisms of written word production: Insights from the written blocked cyclic naming paradigm. Read Writ. 2019 Jan;32(1):65-94. doi: 10.1007/s11145-017-9742-4. Epub 2017 Apr 12. PMID 30686861
- [Background] Ellenblum G, Purcell JJ, Song X, Rapp B. High-level Integrative Networks: A Resting-state fMRI Investigation of Reading and Spelling. J Cogn Neurosci. 2019 Jul;31(7):961-977. doi: 10.1162/jocn_a_01405. Epub 2019 Apr 2. PMID 30938593
- [Background] Rapp B, Wiley RW. Re-learning and remembering in the lesioned brain. Neuropsychologia. 2019 Sep;132:107126. doi: 10.1016/j.neuropsychologia.2019.107126. Epub 2019 Jun 19. PMID 31226267
- [Background] Tao Y, Rapp B. The effects of lesion and treatment-related recovery on functional network modularity in post-stroke dysgraphia. Neuroimage Clin. 2019;23:101865. doi: 10.1016/j.nicl.2019.101865. Epub 2019 May 22. PMID 31146116
- [Background] Wiley RW, Rapp B. From complexity to distinctiveness: The effect of expertise on letter perception. Psychon Bull Rev. 2019 Jun;26(3):974-984. doi: 10.3758/s13423-018-1550-6. PMID 30478777
- [Background] Purcell JJ, Rapp B. Local response heterogeneity indexes experience-based neural differentiation in reading. Neuroimage. 2018 Dec;183:200-211. doi: 10.1016/j.neuroimage.2018.07.063. Epub 2018 Aug 1. PMID 30076891
- [Background] Hepner C, McCloskey M, Rapp B. Do reading and spelling share orthographic representations? Evidence from developmental dysgraphia. Cogn Neuropsychol. 2017 May-Jun;34(3-4):119-143. doi: 10.1080/02643294.2017.1375904. Epub 2017 Sep 21. PMID 28934055
- [Background] McCloskey M, Rapp B. Developmental dysgraphia: An overview and framework for research. Cogn Neuropsychol. 2017 May-Jun;34(3-4):65-82. doi: 10.1080/02643294.2017.1369016. Epub 2017 Sep 14. PMID 28906176
- [Background] Rothlein D, Rapp B. The role of allograph representations in font-invariant letter identification. J Exp Psychol Hum Percept Perform. 2017 Jul;43(7):1411-1429. doi: 10.1037/xhp0000384. Epub 2017 Apr 3. PMID 28368166
- [Background] Breining B, Nozari N, Rapp B. Does segmental overlap help or hurt? Evidence from blocked cyclic naming in spoken and written production. Psychon Bull Rev. 2016 Apr;23(2):500-6. doi: 10.3758/s13423-015-0900-x. PMID 26179140
- [Background] Nozari N, Freund M, Breining B, Rapp B, Gordon B. Cognitive control during selection and repair in word production. Lang Cogn Neurosci. 2016;31(7):886-903. doi: 10.1080/23273798.2016.1157194. Epub 2016 Apr 14. PMID 28133620
- [Background] Wiley RW, Wilson C, Rapp B. The effects of alphabet and expertise on letter perception. J Exp Psychol Hum Percept Perform. 2016 Aug;42(8):1186-203. doi: 10.1037/xhp0000213. Epub 2016 Feb 25. PMID 26913778
- [Background] Rapp B, Purcell J, Hillis AE, Capasso R, Miceli G. Neural bases of orthographic long-term memory and working memory in dysgraphia. Brain. 2016 Feb;139(Pt 2):588-604. doi: 10.1093/brain/awv348. Epub 2015 Dec 17. PMID 26685156
- [Background] Nickels L, Rapp B, Kohnen S. Challenges in the use of treatment to investigate cognition. Cogn Neuropsychol. 2015;32(3-4):91-103. doi: 10.1080/02643294.2015.1056652. PMID 26377505
- [Background] Rapp B, Fischer-Baum S, Miozzo M. Modality and morphology: what we write may not be what we say. Psychol Sci. 2015 Jun;26(6):892-902. doi: 10.1177/0956797615573520. Epub 2015 Apr 29. PMID 25926478
- [Background] Purcell JJ, Shea J, Rapp B. Beyond the visual word form area: the orthography-semantics interface in spelling and reading. Cogn Neuropsychol. 2014;31(5-6):482-510. doi: 10.1080/02643294.2014.909399. Epub 2014 May 16. PMID 24833190
- [Background] Fischer-Baum S, Rapp B. The analysis of perseverations in acquired dysgraphia reveals the internal structure of orthographic representations. Cogn Neuropsychol. 2014;31(3):237-65. doi: 10.1080/02643294.2014.880676. Epub 2014 Feb 5. PMID 24499188
- [Background] Rothlein D, Rapp B. The similarity structure of distributed neural responses reveals the multiple representations of letters. Neuroimage. 2014 Apr 1;89:331-44. doi: 10.1016/j.neuroimage.2013.11.054. Epub 2013 Dec 7. PMID 24321558
- [Background] Tainturier MJ, Bosse ML, Roberts DJ, Valdois S, Rapp B. Lexical neighborhood effects in pseudoword spelling. Front Psychol. 2013 Nov 28;4:862. doi: 10.3389/fpsyg.2013.00862. eCollection 2013. PMID 24348436
- [Background] Purcell JJ, Rapp B. Identifying functional reorganization of spelling networks: an individual peak probability comparison approach. Front Psychol. 2013 Dec 25;4:964. doi: 10.3389/fpsyg.2013.00964. eCollection 2013. PMID 24399981
- [Background] Dufor O, Rapp B. Letter representations in writing: an fMRI adaptation approach. Front Psychol. 2013 Oct 28;4:781. doi: 10.3389/fpsyg.2013.00781. eCollection 2013. PMID 24194724
- [Background] Rapp B, Damian M. (2018). From thought to action: Producing written language. In, Rueschemeyer, S.A & Gaskell, G. (Eds.) Oxford Handbook of Psycholinguistics. Oxford University Press.
- [Background] Nickels L, Kohnen S, Rapp B. (Eds.). (2018). Treatment as a tool for investigating cognition. Psychology Press.
- [Background] Rapp B, Purcell J. (2017). Understanding how we produce written words: Lessons from the brain. In, De Zubicaray, G. and Schiller, N.O. (Eds.) Oxford Handbook of Neurolinguistics. Oxford University Press.
- [Background] Rapp B, Fischer-Baum S. (2014). Representation of orthographic knowledge. In Ferreira, Goldrick and Miozzo (Eds.) Oxford Handbook on Language Production. Oxford University Press.
- [Background] Riley EA, Thompson CK. Training Pseudoword Reading in Acquired Dyslexia: A Phonological Complexity Approach. Aphasiology. 2015 Feb 1;29(2):129-150. doi: 10.1080/02687038.2014.955389. PMID 26085708
- [Background] Lee J, Yoshida M, Thompson CK. Grammatical Planning Units During Real-Time Sentence Production in Speakers With Agrammatic Aphasia and Healthy Speakers. J Speech Lang Hear Res. 2015 Aug;58(4):1182-94. doi: 10.1044/2015_JSLHR-L-14-0250. PMID 25908309
- [Background] Wang H, Thompson CK. Assessing Syntactic Deficits in Chinese Broca's aphasia using the Northwestern Assessment of Verbs and Sentences-Chinese (NAVS-C). Aphasiology. 2016;30(7):815-840. doi: 10.1080/02687038.2015.1111995. Epub 2015 Nov 16. PMID 27453620
- [Background] Cho-Reyes S, Mack JE, Thompson CK. Grammatical Encoding and Learning in Agrammatic Aphasia: Evidence from Structural Priming. J Mem Lang. 2016 Dec;91:202-218. doi: 10.1016/j.jml.2016.02.004. Epub 2016 Mar 21. PMID 28924328
- [Background] Mack JE, Nerantzini M, Thompson CK. Recovery of Sentence Production Processes Following Language Treatment in Aphasia: Evidence from Eyetracking. Front Hum Neurosci. 2017 Mar 13;11:101. doi: 10.3389/fnhum.2017.00101. eCollection 2017. PMID 28348524
- [Background] Mack JE, Thompson CK. Recovery of Online Sentence Processing in Aphasia: Eye Movement Changes Resulting From Treatment of Underlying Forms. J Speech Lang Hear Res. 2017 May 24;60(5):1299-1315. doi: 10.1044/2016_JSLHR-L-16-0108. PMID 28474086
- [Result] Barbieri E, Mack J, Chiappetta B, Europa E, Thompson CK. Recovery of offline and online sentence processing in aphasia: Language and domain-general network neuroplasticity. Cortex. 2019 Nov;120:394-418. doi: 10.1016/j.cortex.2019.06.015. Epub 2019 Jul 13. PMID 31419597
- [Result] Thompson CK, Walenski M, Chen Y, Caplan D, Kiran S, Rapp B, Grunewald K, Nunez M, Zinbarg R, Parrish TB. Intrahemispheric Perfusion in Chronic Stroke-Induced Aphasia. Neural Plast. 2017;2017:2361691. doi: 10.1155/2017/2361691. Epub 2017 Mar 5. PMID 28357141
- [Result] Lukic S, Barbieri E, Wang X, Caplan D, Kiran S, Rapp B, Parrish TB, Thompson CK. Right Hemisphere Grey Matter Volume and Language Functions in Stroke Aphasia. Neural Plast. 2017;2017:5601509. doi: 10.1155/2017/5601509. Epub 2017 May 9. PMID 28573050
- [Result] Lukic S, Thompson CK, Barbieri E, Chiappetta B, Bonakdarpour B, Kiran S, Rapp B, Parrish TB, Caplan D. Common and distinct neural substrates of sentence production and comprehension. Neuroimage. 2021 Jan 1;224:117374. doi: 10.1016/j.neuroimage.2020.117374. Epub 2020 Sep 17. PMID 32949711
- [Result] Higgins J, Barbieri E, Wang X, Mack J, Caplan D, Kiran S, Rapp B, Thompson C, Zinbarg R, Parrish T. Reliability of BOLD signals in chronic stroke-induced aphasia. Eur J Neurosci. 2020 Oct;52(8):3963-3978. doi: 10.1111/ejn.14739. Epub 2020 Apr 28. PMID 32282965
- [Result] Europa E, Gitelman DR, Kiran S, Thompson CK. Neural Connectivity in Syntactic Movement Processing. Front Hum Neurosci. 2019 Feb 13;13:27. doi: 10.3389/fnhum.2019.00027. eCollection 2019. PMID 30814941
- [Result] Lukic S, Meltzer-Asscher A, Higgins J, Parrish TB, Thompson CK. Neurocognitive correlates of category ambiguous verb processing: The single versus dual lexical entry hypotheses. Brain Lang. 2019 Jul;194:65-76. doi: 10.1016/j.bandl.2019.04.005. Epub 2019 May 16. PMID 31103888
- [Result] Hsu CJ, Thompson CK. Manual Versus Automated Narrative Analysis of Agrammatic Production Patterns: The Northwestern Narrative Language Analysis and Computerized Language Analysis. J Speech Lang Hear Res. 2018 Feb 15;61(2):373-385. doi: 10.1044/2017_JSLHR-L-17-0185. PMID 29411008
- [Result] Thompson CK. Single subject controlled experiments in aphasia: the science and the state of the science. J Commun Disord. 2006 Jul-Aug;39(4):266-91. doi: 10.1016/j.jcomdis.2006.02.003. Epub 2006 Apr 25. PMID 16635494
- [Result] Mack JE, Meltzer-Asscher A, Barbieri E, Thompson CK. Neural correlates of processing passive sentences. Brain Sci. 2013 Aug 2;3(3):1198-214. doi: 10.3390/brainsci3031198. PMID 24961525
- [Result] Meltzer-Asscher A, Mack JE, Barbieri E, Thompson CK. How the brain processes different dimensions of argument structure complexity: evidence from fMRI. Brain Lang. 2015 Mar;142:65-75. doi: 10.1016/j.bandl.2014.12.005. Epub 2015 Feb 4. PMID 25658635
- [Result] Schuchard J, Nerantzini M, Thompson CK. Implicit learning and implicit treatment outcomes in individuals with aphasia. Aphasiology. 2017;31(1):25-48. doi: 10.1080/02687038.2016.1147526. Epub 2016 Feb 19. PMID 28603329
- [Result] Mack JE, Wei AZ, Gutierrez S, Thompson CK. Tracking sentence comprehension: Test-retest reliability in people with aphasia and unimpaired adults. J Neurolinguistics. 2016 Nov;40:98-111. doi: 10.1016/j.jneuroling.2016.06.001. Epub 2016 Jun 24. PMID 27867260
- [Result] Schuchard J, Thompson CK. Sequential learning in individuals with agrammatic aphasia: evidence from artificial grammar learning. J Cogn Psychol (Hove). 2017;29(5):521-534. doi: 10.1080/20445911.2017.1293065. Epub 2017 Feb 17. PMID 28690782
- [Derived] Johnson JP, Meier EL, Pan Y, Kiran S. Treatment-related changes in neural activation vary according to treatment response and extent of spared tissue in patients with chronic aphasia. Cortex. 2019 Dec;121:147-168. doi: 10.1016/j.cortex.2019.08.016. Epub 2019 Sep 19. PMID 31627014
- See also: Boston University's Aphasia Research Laboratory — http://www.bu.edu/aphasiaresearch/
- See also: Johns Hopkins University's CogNeuro Research Laboratory — http://sites.krieger.jhu.edu/cogneuro-lab/